CLINICAL TRIAL: NCT05913349
Title: Effectiveness of Group Cognitive Behavioral Therapy for Psychological Sub-health: A Randomized Controlled Trial
Brief Title: Effectiveness of Group Cognitive Behavioral Therapy for Psychological Sub-health
Acronym: EGCBTPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81725005-7
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-04

CONDITIONS: Mental Suffering
Keywords: mental sub-health; Group Cognitive Behavioral Therapy (GCBT); wearable devices; EMA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The clinical response of the group cognitive behavioural therapy (Experimental): A randomized controlled study of GCBT with one-month and six-month post-treatment follow-up was conducted to explore the short- and long-term efficacy of GCBT on mental sub-health
  Interventions: Behavioral: Group Cognitive Behavioral Therapy (GCBT)
- The alterations of behavior and physiological features in the group cognitive behavioral therapy. (Experimental): To understand the possible biological mechanism underlying the efficacy of group cognitive behavioral therapy by analyzing alterations of the alterations of behaviors and Physiological features in the group cognitive behavioral therapy features.
  Interventions: Behavioral: Group Cognitive Behavioral Therapy (GCBT)

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy (GCBT) — Group cognitive behavioral therapy can achieve its therapeutic effect by enhancing emotion regulation and cognitive control, and by improving the activation patterns of the brain's internal networks to promote self-regulation. This can help individuals better manage emotional fluctuations in daily life, resulting in further improvement of depressive and anxious symptoms.

SUMMARY:
Mental health has become an increasing concern, especially since the beginning of the COVID-19 pandemic. However, not all individuals in mental suboptimal states require pharmacological treatment. Cognitive Behavioral Therapy（CBT） can achieve its therapeutic effect by improving activation patterns of the brain's internal networks to promote self-regulation.

The study was designed as a randomized clinical trial with two groups, the GCBT group and the Waiting group, in a state of mental subluxation. the GCBT group received both self-help therapy and on-site guidance, while the Waiting group received the GCBT intervention after treatment in the GCBT group. Data collection was conducted by trained, certified and qualified personnel.

The study was designed to use assessment wearable devices (WD) and mobile apps (MA) for behavioral data and EMA collection during treatment, and the extracted behavioral characteristics were used as objective indicators for long-term and short-term efficacy assessment of GCBT, further understand the possible biological mechanism underlying the efficacy of GCBT by analyzing digital biomarkers.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial designed to assess the efficacy of GCBT compared to a waiting group for mental sub-health. Participants will be randomly (1:1) assigned to the GCBT group and the waiting group. All participants will receive 4 sessions (1 session per week) of 90 minutes each for 4 weeks.The GCBT group will receive cognitive behavioral therapy at the 1st-4th weeks, while the waiting group will receive cognitive behavioral therapy at the 5th-8th weeks. Before GCBT (baseline) and after GCBT (4th weeks, 8th weeks, 28th weeks), both groups will be assessed for clinical symptoms; during the 4 weeks of the intervention, we will collect sensor data and daily diary feedback. The GCBT is mainly divided into four stages, and each stage has a topic. The topic of each stage as follow:# understanding depression, anxiety, and CBT;# understanding automatic thinking and negative automatic thinking;# identifying and correcting negative automatic thinking identification; identifying and correcting intermediate beliefs;#understanding core beliefs and mastering correction techniques.The purposes of the present study are to: 1) evaluate the clinical response the GCBT in mental sub-health. 2) further understand the possible biological mechanism underlying the efficacy of GCBT by analyzing digital biomarkers.

ELIGIBILITY:
Inclusion Criteria:

A total of > 5 on PHQ-9 or a total of > 5 on GAD-7

Exclusion Criteria:

Acute suicidal thoughts, With a severe or potentially confounding psychiatric disorder (e.g. psychosis, substance misuse).

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9; range: 0-27) at 4th weeks, 8th weeks, 28th weeks. | Baseline, 4th weeks, 8th weeks and 28th weeks
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Change from baseline in anxiety symptoms assessed by the Generalized Anxiety Disorder-7 (GAD-7, range: 0-21) at 4th weeks, 8th weeks, 28th weeks. | Baseline, 4th weeks, 8th weeks and 28th weeks
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at 4th weeks, 8th weeks and 28th weeks. | Baseline, 4th weeks, 8th weeks and 28th weeks
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.
Change from baseline in perceived stress assessed by the Perceived Stress Scale-14 (PSS-14; range: 0-56) at 4th weeks, 8th weeks and 28th weeks. | Baseline, 4th weeks, 8th weeks and 28th weeks
  The total scores of these questionnaires were interpreted as follows: normal (0-28), moderate (29-42), severe (43-56).
Change from baseline in suicidal ideation assessed by the Beck Scale for Suicide (BSS-14; range: 0-38) at 4th weeks, 8th weeks and 28th weeks. | Baseline, 4th weeks, 8th weeks and 28th weeks
  The total scores of these questionnaires were interpreted as follows: no or low suicidal ideation (0-8), moderate suicidal ideation(9-16), high suicidal ideation (17-38).

SECONDARY OUTCOMES:
Change from PPG, ACC, heart rate, blood oxygen, sleep time, RRI, step during intervention | During the treatment period
  The sensor data collection time period from 7am to 9pm
Change from daily mood and energy during intervention | At 7am and 9pm daily during the treatment period
  Mood and energy are assessed by a single item each, "On a scale of 1 (very happy) to 7 (very sad), how is your mood right now?" "On a scale of 1 (very tired) to 7 (energetic), how is your energy right now?"

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang Study Chair, PHD, Study Chair — Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Zhou K, Lin Z, Shen H, Liu R, Su Z, Womer FY, Wang Y, Wei Y, Zhu R, Zheng J, Zhang X, Wang F. Evaluation of the efficacy of group cognitive behavioral therapy on anxiety in college students based on wearable devices and mobile applications: a randomized controlled trial. BMC Psychiatry. 2025 Nov 29;26(1):6. doi: 10.1186/s12888-025-07572-y. PMID 41318529
- [Derived] Lin Z, Zheng J, Wang Y, Su Z, Zhu R, Liu R, Wei Y, Zhang X, Wang F. Prediction of the efficacy of group cognitive behavioral therapy using heart rate variability based smart wearable devices: a randomized controlled study. BMC Psychiatry. 2024 Mar 6;24(1):187. doi: 10.1186/s12888-024-05638-x. PMID 38448895